CLINICAL TRIAL: NCT01160432
Title: The Safety and Tolerability of Methadone/Naloxone Combination in Opioid Substitution Treatment
Brief Title: Naloxone Methadone Combination (NAMEKO)
Acronym: NAMEKO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Ulrich Tacke, MD, PhD, docent, Kuopio University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KUH5703433; 2010-021814-43 (EudraCT Number)
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Opiate Dependence
Keywords: opiate dependence; methadone; naloxone; withdrawal symptom; substitution treatment
MeSH Terms: conditions — Opioid-Related Disorders; Substance Withdrawal Syndrome | interventions — Methadone; Naloxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone naloxone combination product 2/0,04 mg/ml (Experimental): Methadone 2 mg/ml in combination with naloxone 0,04 mg/ml
  Interventions: Drug: Methadone, naloxone
- Methadone 2 mg/ml (Active Comparator): Normal treatment except the dilution of methadone solution (5 mg/ml → 2 mg/ml).
  Interventions: Drug: Methadone, naloxone

INTERVENTIONS:
Drug: Methadone, naloxone — Methadone 2 mg/ml in combination with naloxone 0,04 mg/ml daily according to patient's individual dose. At first open label pilot using single (individual) dosage for 2 patients. After that crossover study using methadone 2 mg/ml in combination with naloxone 0,04 mg/ml compared to methadone 2 mg/ml alone in one week's periods for four weeks.
  Other Names: Methadone Martindale Pharma

SUMMARY:
The aim of the study is to examine the tolerability and abuse potential of the diluted methadone solution (5 mg/ml → 2 mg/ml) in combination with naloxone in opioid substitution treatment.

Study hypothesis: Treatment with this diluted combination product is safer than with methadone alone (5 mg/ml) and combination product does not precipitate withdrawal symptoms in opioid dependent patients.

ELIGIBILITY:
Inclusion Criteria:

* opioid dependence
* methadone treatment
* no changes in methadone dose during the last 10 days
* good treatment compliance according to doctor
* normal ALAT and AFOS values (increased if double the normal level)

Exclusion Criteria:

* severe renal or hepatic failure
* acute psychosis
* age under 18
* pregnancy
* legal incompetence
* severe somatic disease
* chaotic situation in life
* medication or disease which is contraindication to study treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Withdrawal symptoms (Clinical Opioid Withdrawal Scale COWS, Subjective Opiate Withdrawal Scale SOWS) | 1/2 hours after the first intake of medicine every week
  COWS is completed by the nurse and SOWS by the patient. Withdrawal symptoms are estimated every week after the intake of new product (blinded).

SECONDARY OUTCOMES:
The effectiveness of treatment (Treatment Outcomes Profile TOP) | Before study begins, after 4 week study period and 4 weeks after the end of the clinical phase.
  Structured interview designed to measure the effectiveness and outcomes of opioid substitution treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Tacke, MD, PhD, Study Director — Kuopio University Hospital, University of Eastern Finland
Locations (1):
- Kuopio University Hospital, Kuopio, Finland